CLINICAL TRIAL: NCT01879072
Title: Prospective Multi-Center Cohort for the Evaluation of Biomarkers Predicting Risk of Complications and Mortality Following Allogeneic HCT (BMT CTN #1202)
Brief Title: Prospective Cohort for the Evaluation of Biomarkers Following HCT (BMT CTN 1202)
Status: Completed | Type: Observational
Sponsor: Medical College of Wisconsin (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); National Cancer Institute (NCI) (NIH); Blood and Marrow Transplant Clinical Trials Network (Network); National Marrow Donor Program (Other)
Responsible Party: Sponsor
Other Study IDs: BMTCTN1202; U10HL069294-11 (NIH); 5U24CA076518 (NIH)
Record Dates: First submitted 2013-06-11; First posted 2013-06-17 (Estimated); Results first posted 2018-05-29 (Actual); Last update posted 2022-12-09 (Actual); Status verified 2022-12

CONDITIONS: Allogeneic Hematopoietic Stem Cell Transplantation
Keywords: Biomarkers; Hematopoietic stem cell transplant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — 10mL serum for Proteomic studies for patients at the following time points: pre-transplant, days 7, 14, 21, 28, 42, 56, and 90.
  Gene Expression studies will include the following:
  * PAXgene Lysates-source whole blood RNA (15 ml blood) for 240 patients collected on days 21, 56, and 90.
  * CytoChex tube for Immunophenotyping (4-5 mL blood) collected on days 21, 56, and 90.
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The goal of this protocol is to establish a cohort of at least 1500 biologic samples collected prospectively from patients treated in BMT CTN centers that will be a shared bio specimen resource for conducting future allogeneic hematopoietic stem cell transplantation (HCT) correlative studies.

DETAILED DESCRIPTION:
The goal of this protocol is to establish a cohort of biologic samples collected prospectively from patients treated in BMT CTN centers that will be a shared bio specimen resource for conducting future allogeneic HCT correlative studies. This resource is designed to allow genomic, proteomic and transcriptional data to be integrated with high quality clinical phenotype and outcomes data to identify risk factors for development and severity of acute GVHD, chronic GVHD, organ toxicity, relapse, mortality, infection and other clinically significant complications occurring after allogeneic HCT.

To achieve this goal, patients and donors will be recruited and consent obtained at the time that they enroll on BMT CTN protocols where enrollment occurs at or before transplantation or prior to start of conditioning for patients enrolled on non-BMT CTN studies or treated as standard of care. Samples will be collected: (1) from patients and donors pre-transplant; and, (2) from patients post-transplant on a calendar schedule through the first 3 months post-HCT. For patients co-enrolled on BMT CTN studies, clinical data will be collected in the context of the primary transplant protocols. For patients not enrolled on BMT CTN protocols, clinical data on early post-transplant events will be collected using the same data collection forms and systems that are used on BMT CTN trials. Additional clinical data for both BMT CTN and non-BMT CTN patients will be available from data submitted to the Center for International Blood and Marrow Transplant Research (CIBMTR) using the CIBMTR Comprehensive Report Forms. This protocol also leverages ongoing pre-transplant donor-recipient sample collection performed by the CIBMTR and National Marrow Donor Program (NMDP). Success in establishing this shared resource will inspire future investigator initiated research proposals and will allow investigators to take advantage of National Institutes of Health (NIH) funding initiatives.

ELIGIBILITY:
Inclusion Criteria:

1. Recipients of first allogeneic hematopoietic cell transplants that are transplanted in U.S. centers that participate in the NMDP/CIBMTR's "Protocol for a Research Sample Repository for Allogeneic Hematopoietic Stem Cell Transplantation and Marrow Toxic Injuries" and receive a cord blood graft or receive a bone marrow or peripheral blood graft from a related donor or from an unrelated donor in an NMDP-affiliated Donor Center or Registry participating in that same protocol.

   This transplant and donor center restriction is to allow linkage with pretransplant donor specimens collected under the NMDP/CIBMTR protocol. Current data indicate that >90% of donors approached under this protocol agree to provide samples
2. Patients with any malignant or non-malignant hematologic disorder will be eligible for enrollment on this protocol. A subset of 240 sequential patients with acute leukemia in first or second remission will also provide research samples for gene expression studies.
3. Children may participate in this study but must weigh at least 20 kilograms given the volume (100ml) and number of blood draws during this study. Subjects must weigh at least 30 kg to provide research samples for gene expression studies (additional 40 ml).
4. All participants or parent/legal guardian must sign an informed consent for this study.

Because studies using this resource will require linking with clinical data collected by CIBMTR, all participants or parent/legal guardian must also consent to participate in "Protocol for a Research Database for Hematopoietic Cell Transplantation and Marrow Toxic Injuries".

Exclusion Criteria:

* N/A

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All U.S. Allogeneic Transplant Donors and Recipients weighing 20 or more kg may participate in the collection of samples.
Sampling Method: Non-Probability Sample
Enrollment: 1860 (Actual)
Dates: Start 2013-06 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary Horowitz, MD, MS, Study Director — Center for International Blood and Marrow Transplant Research (CIBMTR), Medical College of Wisconsin
Locations (42):
- United States (42):
  - Phoenix Children's Hospital, Phoenix, Arizona
  - City of Hope National Medical Center, Duarte, California
  - Children's Hospital at Oakland, Oakland, California
  - University of CA, SF, San Francisco, California
  - Stanford Hospitals and Clinics, Stanford, California
  - Nemours/Alfred I. duPont Hospital for Children, Wilmington, Delaware
  - Children's National Medical Center, Washington D.C., District of Columbia
  - University of Florida College of Medicine (Shands), Gainesville, Florida
  - All Children's Hospital, St. Petersburg, Florida
  - H. Lee Moffitt Cancer Center, Tampa, Florida
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Emory University, Atlanta, Georgia
  - BMT at Northside Hospital, Atlanta, Georgia
  - Ann and Robert H. Lurie Children's Hospital, Chicago, Illinois
  - University of Kansas Hospital, Kansas City, Kansas
  - Johns Hopkins, Baltimore, Maryland
  - DFCI/Brigham & Women's, Boston, Massachusetts
  - University of Michigan Medical Center, Ann Arbor, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic - Rochester, Rochester, Minnesota
  - Washington University/Barnes Jewish Hospital, St Louis, Missouri
  - Washington University/St. Louis Children's Hospital, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Roswell Park, Buffalo, New York
  - Mount Sinai Medical Center, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - University of North Carolina Hospital at Chapel Hill, Chapel Hill, North Carolina
  - Duke University, Durham, North Carolina
  - University Hospitals of Cleveland/Case Western, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State/Arthur G. James Cancer Hospital, Columbus, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - University of Pennsylvania Cancer Center, Philadelphia, Pennsylvania
  - Children's Medical Center of Dallas, Dallas, Texas
  - Cook Children's Hospital, Fort Worth, Texas
  - Baylor College of Medicine/The Methodist Hospital, Houston, Texas
  - University of Texas/MD Anderson CRC, Houston, Texas
  - Texas Transplant Institute, San Antonio, Texas
  - Utah BMT/Primary Children's Medical Center, Salt Lake City, Utah
  - Virginia Commonwealth University, Richmond, Virginia
  - Fred Hutchinson Cancer Research Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
Findings will be published in a manuscript.
Time Frame: Within 6 months of official study closure at participating sites.
Access Criteria: Available to the public.
URL: https://biolincc.nhlbi.nih.gov/home/

REFERENCES:
- [Derived] Bhasin-Chhabra B, Wang T, Levine JE, Shenoy S, Perales MA, Bashey A, Raff H, Saber W. Soluble urokinase plasminogen activator receptor and acute kidney injury in hematopoietic cell transplantation. Blood Adv. 2025 Dec 23;9(24):6394-6401. doi: 10.1182/bloodadvances.2025016655. PMID 40991367

RESULTS

PARTICIPANT FLOW:
Groups:
- Allogeneic Hematopoietic Stem Cell Transplant: Participants received allogeneic hematopoietic stem cell transplantation
Period: Overall Study
Arm/Group | Allogeneic Hematopoietic Stem Cell Transplant
Started | 1860
Completed | 1709
Not Completed | 151
Not completed — Withdrawal by Subject | 121
Not completed — Not Transplanted | 30

BASELINE CHARACTERISTICS:
Arm/Group | Allogeneic Hematopoietic Stem Cell Transplant
Number analyzed (Participants) | 1709
Age, Continuous [Median (Full Range); unit: years] | 52.7 [0.5 to 77.3]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 701
  Male | 1008
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 128
  Not Hispanic or Latino | 1552
  Unknown or Not Reported | 29
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 9
  Asian | 59
  Native Hawaiian or Other Pacific Islander | 5
  Black or African American | 203
  White | 1370
  More than one race | 13
  Unknown or Not Reported | 50

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Providing Biologic Samples
Description: The primary outcome will be measured by the number of participants who supply biologic samples. The prospectively collected samples will be a shared bio specimen resource for conducting future correlative studies.
Time Frame: Two years from hematopoietic stem cell transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Allogeneic Hematopoietic Stem Cell Transplant
Number analyzed (Participants) | 1709
Participants | 1709

ADVERSE EVENTS:
Time Frame: Two years post-transplant
Arm/Group | Hematopoietic Stem Cell Transplant
Serious Adverse Events (participants affected / at risk) | 0/1709
Other Adverse Events (participants affected / at risk) | 0/1709

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2015-03-17): https://cdn.clinicaltrials.gov/large-docs/72/NCT01879072/Prot_SAP_ICF_000.pdf